CLINICAL TRIAL: NCT04469218
Title: Dislodgement Infiltration Phlebitis Prevention Eliminating Restarts (DIPPER)
Brief Title: A Clinical Trial Using a New Medical Device to Evaluate Its Impact on IV Care and Clinical Complications
Acronym: DIPPER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lineus Medical (Industry)
Collaborators: Hartford HealthCare (Other); Hartford Hospital (Other); Technomics Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P002
Record Dates: First submitted 2020-07-08; First posted 2020-07-13 (Actual); Results first posted 2024-01-16 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2023-12

CONDITIONS: IV Catheter-Related Infection or Complication
Keywords: IV Care; IV Complication

STUDY DESIGN:
Intervention Model Description: A randomized clinical trial with a control group receiving the standard of care peripheral IV treatment and a second group that utilizes SafeBreak Vascular, a break-away connector, in the peripheral IV.
Masking Description: The use of devices is randomly assigned to subjects in the study, but it is not possible to blind the patient, the care providers, the investigators or the outcomes assessor as to which group received the study device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control Group (No Intervention): Subjects in the control group will receive the standard of care intervention for peripheral IVs at the study hospital.
- SafeBreak Vascular Group (Experimental): Subjects in the SafeBreak Vascular group will have as near to identical treatment as possible to the control group with the exception that a SafeBreak Vascular device will be placed in the peripheral IV line.
  Interventions: Device: SafeBreak Vascular

INTERVENTIONS:
Device: SafeBreak Vascular — SafeBreak Vascular is a breakaway connector that screws into peripheral IV lines using luer connectors on each end. The device is designed to separate when a harmful force is placed on an IV line. Upon separation, valves on each side of the device close. On the patient side of the device, the valve closes to prevent the loss of blood and on the IV pump side of the device, the valve closes to stop the flow of medication. The valve closing on the IV pump side of the line causes the pump's occlusion alarm to sound and notify nurses that the IV needs attention. The nurse is able to throw away the separated SafeBreak Vascular, install a new SafeBreak, and restart the patient's infusion without the negative cascade of events that can occur when a peripheral IV fails.
  Other Names: Patient safety disconnect
  Arms: SafeBreak Vascular Group

SUMMARY:
A clinical trial comparing two groups of patients that are randomized into one group having SafeBreak Vascular attached to their peripheral IV lines and a second control group that receives the current standard of care (no SafeBreak Vascular) to determine SafeBreak Vascular's impact on IV clinical care and complications.

DETAILED DESCRIPTION:
This randomized clinical trial's goal is to determine SafeBreak Vascular's impact, a break-away connector that separates when a harmful force is placed on a peripheral IV line, on IV clinical care and complications.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted into the participating hospital units
* Patients of any gender may participate
* Participants able to provide informed consent or have a legally authorized representative immediately available to provide informed consent
* Patients must have peripheral IV catheter access or need and are planned to have peripheral IV catheter access placed that is anticipated to last a minimum of 24 hours.
* Patients must be receiving intermittent or continuous infusion or have immediate plans to begin an intermittent or continuous infusion
* The patients must be at least 18 years of age with no upper age limit

Exclusion Criteria:

* Unable to obtain informed consent or without an available Legally Authorized Representative or Next of Kin to provide surrogate informed consent
* Age less than or equal to 17
* Patient on comfort care only
* Predicted to have an IV infusion that lasts less than 24 hours
* Patient admitted from the Emergency Department refuses to have new peripheral IV catheter placed by IV team
* Patient has two or more peripheral IV catheters at the same time
* Patient enrolled in a subject drug or device study at the time of enrollment
* Investigator discretion that patient is not suitable for the study
* Patient is COVID-19 positive
* Patient is receiving an IV infusion with gravity tubing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2020-07-14 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee Steere, Principal Investigator — Hartford Hospital
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Group | SafeBreak Vascular Group
Started | 74 | 74
Completed | 69 | 70
Not Completed | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | SafeBreak Vascular Group | Total
Number analyzed (Participants) | 69 | 70 | 139
Age, Continuous [Mean (Full Range); unit: Years] | 59 [24 to 90] | 59 [21 to 89] | 59 [21 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 27 | 59
  Male | 37 | 43 | 80
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 10 | 28
  Not Hispanic or Latino | 51 | 60 | 111
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 10 | 18
  White | 61 | 59 | 120
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Delay in Therapy
Description: A comparison in delays in therapy between the control group and the intervention group.
Time Frame: Patients evaluated at every IV check from time of enrollment to time of discontinuation of IV therapy or up to 7 days, whichever occurs first
Population: All patients in Per Protocol population
Measure: Mean (Standard Deviation); unit: min per 24 hours
Arm/Group | Control Group | SafeBreak Vascular Group
Number analyzed (Participants) | 69 | 70
min per 24 hours | 11.73 (36.56) | 10.89 (41.45)

2. Secondary Outcome: Estimate the Impact for Other Peripheral IV Complications.
Description: A comparison in IV complications (dislodgement, infiltration, and phlebitis VIP =2 or greater) requiring IV restart between the control group and the intervention group.
Time Frame: as for outcome 1
Population: All patients in Per Protocol population
Measure: Number; unit: mechanical complications
Arm/Group | Control Group | SafeBreak Vascular Group
Number analyzed (Participants) | 69 | 70
mechanical complications | 25 | 15

ADVERSE EVENTS:
Time Frame: Patients evaluated and adverse events documents at every IV check from time of enrollment to time of discontinuation of IV therapy or up to 7 days, whichever occurs first
Arm/Group | Control Group | SafeBreak Vascular Group
All-Cause Mortality (participants affected / at risk) | 0/69 | 0/70
Serious Adverse Events (participants affected / at risk) | 2/69 | 2/70
Other Adverse Events (participants affected / at risk) | 33/69 | 26/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=69) | SafeBreak Vascular Group (N=70)
Chest Pain (Cardiac disorders) | 2 (2) | 1 (1)
Unwitnessed Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=69) | SafeBreak Vascular Group (N=70)
Dislodgement (Surgical and medical procedures) | 3 (4) | 2 (2)
Infiltration (Surgical and medical procedures) | 7 (10) | 8 (8)
Phlebitis VIP =/>2 (Surgical and medical procedures) | 10 (10) | 1 (1)
Occlusion (Surgical and medical procedures) | 1 (1) | 4 (4)
Device Crack/Leak (Product Issues) | 0 (0) | 2 (2)
IV Site Bleeding/Fluid Leakage (Surgical and medical procedures) | 1 (1) | 2 (2) — IV Repaced; IV site bleeding or fluid
Mental Status Change/Unwitnessed Fall (Psychiatric disorders) | 3 (5) | 1 (1) — Altered mental status; Confusion, Hallucinations, unresponsive, unwitnessed fall
Blood Chemistry Abnormalities (Blood and lymphatic system disorders) | 7 (8) | 2 (2) — Decreasing hemoglobin&Hematocrit; high/low BP; low platelet count; low potassium; low sodium; O2 desaturation
Skin Reactions (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) — Extremity itching; rash
Pains (General disorders) | 13 (13) | 4 (6) — Abdominal pain; back pain; body aches, lower extremity pain; upper extremity pain; headache
Cardiovascular (Cardiac disorders) | 2 (2) | 4 (4) — Chest pain, shortness of breath
Nausea/Diarrhea (General disorders) | 4 (7) | 2 (3)
Elevated Temperature (General disorders) | 5 (6) | 0 (0)
Urinary Catheter Placed (Renal and urinary disorders) | 1 (1) | 0 (0)
Post-op Complication (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-10-13): https://cdn.clinicaltrials.gov/large-docs/18/NCT04469218/Prot_002.pdf
  • Statistical Analysis Plan (2020-10-13): https://cdn.clinicaltrials.gov/large-docs/18/NCT04469218/SAP_003.pdf
  • Informed Consent Form (2020-07-27): https://cdn.clinicaltrials.gov/large-docs/18/NCT04469218/ICF_001.pdf